CLINICAL TRIAL: NCT01600300
Title: A Double-Blind, Placebo-Controlled Feasibility Study to Evaluate the Efficacy of TESMAC™ (Transcutaneous Electrical Stimulation of the Macula)
Brief Title: Efficacy of Electrical Micro-current Retinal Stimulation for Treatment of Dry Age-related Macular Degeneration
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Acuity Medical International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TESMAC-2002.2
Record Dates: First submitted 2012-05-14; First posted 2012-05-17 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Macular Degeneration
Keywords: Age-related macular degeneration; electrical stimulation; randomized; double blind
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Sham (Placebo Comparator): Treatment with inactivate Tesmac device
  Interventions: Device: Sham Tesmac device
- Tesmac (Active Comparator): Treatment with active Tesmac device
  Interventions: Device: Tesmac

INTERVENTIONS:
Device: Tesmac — Subjects were treated twice daily for five consecutive days, followed by two days untreated, and then treated twice daily for five more consecutive days.
  Other Names: Theramac
  Arms: Tesmac
Device: Sham Tesmac device — Treatment with inactivated Tesmac device on the same schedule as the group treated with the active Tesmac device.
  Arms: Sham

SUMMARY:
Hypothesis: external electrical stimulation of the retina with low level electrical currents improves visual acuity in subjects with age-related dry macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Macular Degeneration, i.e., at least three, hard or soft drusen must be present there must be RPE changes (migration, clumping or atrophy) within the central 6mm of the retina.
2. As a prerequisite for entry into the study, all patients will have their diagnosis of dry AMD confirmed by an ophthalmologist via a retinal exam and Fluorescein Angiography will also determine whether or not the subject is a candidate for laser surgery. Only subjects who have AMD will be admitted to the study.
3. Both sexes are eligible.
4. The best-corrected visual acuity can be no better than 20/40 and no worse than 20/100 in the treated eyes.
5. Age greater than 50.
6. Subjects must be highly motivated, alert, oriented, mentally competent and able to understand and comply with the requirements of the study, abide by the restrictions, return for all required visits, and provide voluntary informed consent.
7. Both eyes of the subject must show no evidence of wet AMD. If one eye is wet and the fellow eye is dry, the subject will be excluded.

Exclusion Criteria:

1. Subjects with seizure disorders.
2. Subjects with additional eye-related diseases that have associated ongoing retinal bleeding.
3. Subjects with any implanted electrical device.
4. Subjects who have smoked, on average, more than half a pack of cigarettes per day during the last 5 years.
5. Subjects with known allergy to contrast dye.
6. Subjects who are in poor general health, have unstable diseases, are terminally ill, have a life expectancy of less than 12 months, are non-ambulatory or bedridden, live in a geographical location which would likely prevent regular attendance at study visits or are considered not suitable for participation by the investigator.
7. Subjects exposed to an investigational device or drug within the past 30 days or involved concurrently in other treatment clinical trials. Note: Subjects participating in studies investigating the natural progression of AMD may not participate in this trial.
8. Subjects unwilling to adhere to visit or examination schedules as described in the study protocol.
9. Subjects with a known history of alcoholism, drug abuse, psychosis, clinical evidence of depression, poor motivation, emotional or intellectual problems, or any other conditions which would likely limit validity of consent or appropriate responses to participate in the study or who are deemed unsuitable psychologically or physiologically for study participation by the investigator.
10. Any subject experiencing an acute stressor that, in the opinion of the investigator, might affect the course or treatment of AMD.
11. Anyone with diagnosis of malignant or poorly controlled glaucoma in the eye(s) that would be treated.
12. Anyone with diabetic retinopathy.
13. Anyone with a progressive corneal dystrophy in the eye(s) that would be treated.
14. Anyone with any noted chorio retinal disease (other than AMD) in the eye(s) that would be treated.
15. Anyone with a progressive nuclear cataract in the eye(s) that would be treated. Stable cortical cataract patients may be included. Any patient with an immature cataract, one in which scattered opacities are separated by clear zones, may be included in the study. All patients with mature, hypermature or morgagnian cataracts in the eye(s) that would be treated will be excluded. Patients with a grade 3 or grade 4 cataract in the eye(s) that would be treated will be excluded. Grade 1 and Grade 2 cataract patients may be included in this study.
16. Subjects participating in an AMD natural history study.
17. Subjects with one eye diagnosed with wet AMD.
18. Subjects with any previous retinal bleeding, injury, or retinal surgery.
19. Subjects that have previously been diagnosed with amblyopia.
20. Subjects currently taking blood-thinning medication.
21. Subjects cannot have previously been involved in a TESMAC™ study.
22. Subjects that take two or more of the following antioxidants daily at the following doses: 500 milligrams of vitamin C; 400 international units of vitamin E; 15 milligrams of beta-carotene; 80 milligrams of zinc as zinc oxide; and two milligrams of copper as cupric oxide and have done this for more than 2 years. These subjects may be included, but their study results will be analyzed separately.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2002-08; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Change in visual acuity | Day 5, Day 12
  Change in visual acuity as measured with ETDRS eye chart

CONTACTS AND LOCATIONS:
Overall Officials: Richard Beauchemin, MD, Principal Investigator — WNC Eye Care Associates PA